CLINICAL TRIAL: NCT05364164
Title: A Phase I, Randomized, Open-Label, Single-Dose, Crossover Study to Evaluate Food Effect on the Pharmacokinetics and Safety of CT-L01 After Oral Administration in Healthy Volunteers
Brief Title: A Food Effect Study of CT-L01 After Oral Administration in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celltrion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CT-L01-103
Record Dates: First submitted 2022-04-19; First posted 2022-05-06 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CT-L01 12.5/1,000 mg FDC Tablet, dosing under fasting condition (Experimental): Alogliptin Benzoate 12.5 mg/Metformin HCl XR 1,000 mg, FDC Tablet, dosing under fasting condition
  Interventions: Drug: CT-L01 12.5/1,000 mg
- CT-L01 12.5/1,000 mg FDC Tablet, dosing under fed condition (Experimental): Alogliptin Benzoate 12.5 mg/Metformin HCl XR 1,000 mg, FDC Tablet, dosing after high-fat meal
  Interventions: Drug: CT-L01 12.5/1,000 mg

INTERVENTIONS:
Drug: CT-L01 12.5/1,000 mg — FDC tablet, 2 tablets at a time, oral administration, dosing under fasting condition
  Arms: CT-L01 12.5/1,000 mg FDC Tablet, dosing under fasting condition
Drug: CT-L01 12.5/1,000 mg — FDC tablet, 2 tablets at a time, oral administration, dosing after high-fat meal
  Arms: CT-L01 12.5/1,000 mg FDC Tablet, dosing under fed condition

SUMMARY:
This is a phase 1, randomized, open-label, single-dose, crossover, single-center study to evaluate food effect on the pharmacokinetics and safety of CT-L01 after oral administration in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subject aged 19 to 50 years, at screening
* A subject who weighs 50 kg or more at the screening visit and has a body mass index (BMI) of 18.0~30.0 kg/m2
* A subject who is judged to be eligible to participate by the results of screening tests (vital signs, clinical laboratory tests, 12-lead ECG, etc.) by the principal investigator within 28 days before the first administration of the investigational drug
* A subject and their partner who agree to use a medically appropriate method of contraception to exclude potential of pregnancy and not to provide sperm or ova from the first dose to 28 days after the last dose of the investigational drug
* A subject who voluntarily signs the consent form after hearing and understanding the purpose and content of this study, thge characteristics of the investigational drugs, expected adverse reactions, and etc.

Exclusion Criteria:

* A subject who has a history or present symptoms of clinically significant liver, kidney, nervous system, respiratory system, digestive system, endocrine system, blood/tumor, urinary system, cardiovascular system, musculoskeletal disease, or psychiatric disease
* A subject who has an acute illness within 28 days prior to the first dose of investigational drug
* A subject who has a history of gastrointestinal surgery that may affect drug absorption (except simple appendectomy or hernia surgery) or has gastrointestinal diseases
* A subject who has taken drugs that induce or inhibit drug metabolizing enzymes such as barbiturates within 1 month prior to the first administration
* A subject who has participated in other clinical trials or bioequivalence studies within 6 months prior to the first dose of the investigational drug
* A subject who is judged unsuitable to participate in this study by the principal investigator

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-07-09 (Actual); Primary Completion 2022-07-19 (Actual); Study Completion 2022-07-25 (Actual)

PRIMARY OUTCOMES:
AUClast (Area under the plasma concentration-time curve) | Pre-dose(0.00), 0.25, 0.50, 1.00, 1.50, 2.00, 2.50, 3.00, 4.00, 5.00, 6.00, 7.00, 8.00, 10.00, 12.00, 16.00, 24.00, 36.00, 48.00, and 72.00 hours
Cmax (Peak Plasma Concentration) | Pre-dose(0.00), 0.25, 0.50, 1.00, 1.50, 2.00, 2.50, 3.00, 4.00, 5.00, 6.00, 7.00, 8.00, 10.00, 12.00, 16.00, 24.00, 36.00, 48.00, and 72.00 hours

SECONDARY OUTCOMES:
AUCinf (Area under the plasma concentration-time curve from time 0 to infinity) | Pre-dose(0.00), 0.25, 0.50, 1.00, 1.50, 2.00, 2.50, 3.00, 4.00, 5.00, 6.00, 7.00, 8.00, 10.00, 12.00, 16.00, 24.00, 36.00, 48.00, and 72.00 hours
AUClast/AUCinf | Pre-dose(0.00), 0.25, 0.50, 1.00, 1.50, 2.00, 2.50, 3.00, 4.00, 5.00, 6.00, 7.00, 8.00, 10.00, 12.00, 16.00, 24.00, 36.00, 48.00, and 72.00 hours
Tmax (Time of peak plasma concentration) | Pre-dose(0.00), 0.25, 0.50, 1.00, 1.50, 2.00, 2.50, 3.00, 4.00, 5.00, 6.00, 7.00, 8.00, 10.00, 12.00, 16.00, 24.00, 36.00, 48.00, and 72.00 hours
t1/2 (Half-life) | Pre-dose(0.00), 0.25, 0.50, 1.00, 1.50, 2.00, 2.50, 3.00, 4.00, 5.00, 6.00, 7.00, 8.00, 10.00, 12.00, 16.00, 24.00, 36.00, 48.00, and 72.00 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Chungnam National University Hospital, Daejeon, South Korea